CLINICAL TRIAL: NCT03411616
Title: Eating Behavior, Food Craving and Relation to Excessive Weight Gain in Patients Submitted to Liver Transplantation
Status: Completed | Type: Observational
Sponsor: Federal University of Minas Gerais (Other)
Collaborators: Coordenação de Aperfeiçoamento de Pessoal de Nível Superior. (Other Government); Conselho Nacional de Desenvolvimento Científico e Tecnológico (Other Government)
Responsible Party: Principal Investigator, Maria Isabel Toulson Davisson Correia, Professor, Federal University of Minas Gerais
Other Study IDs: CAAE - 10726313.3.0000.5149
Record Dates: First submitted 2018-01-06; First posted 2018-01-26 (Actual); Last update posted 2018-01-26 (Actual); Status verified 2018-01

CONDITIONS: Eating Behavior; Liver Transplant
Keywords: Eating behavior; Excessive weight; Food craving; Liver transplantation; Obesity; Weight gain
MeSH Terms: conditions — Feeding Behavior; Obesity; Weight Gain

STUDY DESIGN:
Observational Model: Other | Time Perspective: Cross-Sectional
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Excessive weight gain, obesity and metabolic syndrome are highly prevalent in patients undergoing liver transplantation. Traditional methods of assessing dietary intake have failed to demonstrate an association between these problems and dietary intake. Patients with an indication for transplantation due to ethanolic cirrhosis, ex-smokers and those with a previous history of overweight were identified as being at greater risk for overweight and metabolic syndrome, and these factors may be related to the change in eating behavior after the operation. Objective: To evaluate the eating behavior, the occurrence of food craving and relation to weight gain, overweight and obesity after liver transplantation. Method: This is a cross-sectional study in which adult and elderly patients in follow-up at the Hepatic Transplant Outpatient Clinic of the Alpha Institute of Gastroenterology of the Federal University of Minas Gerais were evaluated for eating behavior and food craving. The evaluation of the eating behavior was performed with the help of the Three Factor Eating Questionnaire-R21 (TFEQ-R21), translated version and validated for Portuguese. Food Craving Questionnaires State (FCQ-S) and Trait (FCQ-T) and the Brazilian Inventory of Foods Related to Craving (FCI-Br) were used in the translated and validated versions for Portuguese. Demographic, lifestyle, clinical and anthropometric variables of the evaluated patients were obtained through electronic medical records. Weight gain was assessed by the difference between the current weight and the first post-transplant outpatient weight.

ELIGIBILITY:
Inclusion Criteria:

* Patients who undergone liver transplantation
* At least 18 years of age
* Patients regularly followed up at the Bias Fortes outpatient clinic
* Patients who agreed to participate in the study

Exclusion Criteria:

* Patients who were unable to write and who did not have an accompanying person present as a literate person
* Pregnant or nursing women

Min Age: 18 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: Patients who undergone liver transplantation at least 18 years of age, who were regularly followed up at the Bias Fortes outpatient clinic
Sampling Method: Non-Probability Sample
Enrollment: 301 (Actual)
Dates: Start 2016-08-23 (Actual); Primary Completion 2017-02-23 (Actual); Study Completion 2017-02-23 (Actual)

PRIMARY OUTCOMES:
Eating behavior | 40 minutes
  The evaluation of the eating behavior was performed with the help of the Three Factor Eating Questionnaire-R21 (TFEQ-R21), translated version and validated for Portuguese. This is a self-report questionnaire composed of 21 items, with 4 response options for questions 1 to 20 and question 21 is evaluated on a likert 8-point scale. TFEQ-R21 evaluates 3 types of eating behavior: cognitive restriction (CR), emotional eating (EE) and uncontrolled eating (UE). The CR scale assesses the tendency to control food intake in order to influence body weight and body shape, with 6 items in scale. The EE scale measures the propensity to overeat in relation to negative mood states, e.g., when feeling lonely, anxious, or depressed, has 6 items. The UE scale assesses the tendency to lose control over eating when feeling hungry or when exposed to external stimuli, has 9 of items in scale. Each score ranges from 0 to 100, with higher score indicative of greater level in the eating behavior of interest.

SECONDARY OUTCOMES:
Food Craving Questionnaires State (FCQ-S) | 20 minutes
  The FCQ-State consists of 15 questions, grouped into five dimensions: An intense desire to eat (Desire); anticipation of positive reinforcement that may result from eating (Pos R); anticipation of relief from negative states and feelings as a result of eating (Neg R); thoughts of preoccupation with food and lack of control over eating (Lack Co); and craving as part of the sensation of hunger, a physiological state (Hunger). Participants must answer each question related to what they are feeling at the moment, using a Likert scale of five points, the extremes of which are "(1) strongly disagree" and "(5) strongly agree". The full-scale score corresponds to the sum of the scores obtained in each dimension, which is calculated by simply adding them. Total scores can vary from 15 to 75.
Food Craving Questionnaires Trait (FCQ-T) | 20 minutes
  consume food (Plan); environmental cues that may trigger food craving (Environ); thoughts or preoccupation with food (Thoughts); craving as a physiological state (Hunger); possible lack of control over eating if food is being eaten (Lack Co); emotions that may be experienced before or during food cravings or eating (Emotion); and guilt that may be experienced because of cravings and/or giving in to them (Guilt). The answers are recorded on a Likert scale, ranging from "(1) never or not applicable" to "(6) Always," referring to the frequency with each statement applies to the participant. Full-scale and factor-scale totals are obtained by the sum of the corresponding item scores. Thus, the overall score can range from 39 to 234.
Brazilian Inventory of Foods Related to Craving (FCI-Br) | 20 minutes
  The Brazilian Inventory of Foods Related to Craving (FCI-Br) begins with a short definition of food cravings behavior, followed by the question ''Over the past month, how often have you experienced a craving for the food listed below?''. Each of the foods listed was evaluated using a five point Likert scale ranging from: "(1) never" to "(5) almost every day". The total score of each FCI-Br subscale was calculated by adding the scores obtained for each item that comprised it.

OTHER OUTCOMES:
Demographic, lifestyle, clinical and anthropometric variables | 40 minutes
  Own Checklist - Demographic variables as well as habitual life style, clinical and anthropometric characteristics were assessed. Clinical variables encompassed indication for LTx, time since LTx and current immunossupressive drugs. Self reported current and past smoking and alcohol consumption were also collected. The patients' weight (kilograms) on the first outpatient visit after LTx was collected from their medical recorders, it is regularly measured with patients wearing light street clothing, no shoes, on a calibrated mechanical scale (Filizola®). Current height (meters) and weight (kilograms) of patients were measured on the day of the interview. Considering these weights, weight gain was assessed by the difference between the current weight and the first post-LTx outpatient weight. Nutritional status was defined according to body mass index (BMI) values as underweight, BMI <18.5 kg/m²; normal weight, BMI 18.5-24.9 kg/m²; overweight, BMI 24.9-29.9 kg/m² and obese, BMI >30 kg/m².

CONTACTS AND LOCATIONS:
Locations (1):
- Hospital of Clinics of the University Federal of Minas Gerais, Belo Horizonte, Minas Gerais, Brazil